CLINICAL TRIAL: NCT05518708
Title: A Phase I Single-blind, Randomised, Placebo-controlled, Parallelgroup Design Trial to Investigate the Safety, Tolerability, Pharmacokinetics and Harmacodynamics of Single Rising Doses of BI 3032950 Administered as Intravenous Infusion (Part A) or Subcutaneous Injection (Part B) to Healthy Male Subjects
Brief Title: A Study in Healthy Men to Test How Different Doses of BI 3032950 Are Tolerated
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1486-0001; 2022-002161-15 (EudraCT Number)
Record Dates: First submitted 2022-08-25; First posted 2022-08-29 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BI 3032950 treatment group - part A (Experimental)
  Interventions: Drug: BI 3032950
- BI 3032950 treatment group - part B (Experimental)
  Interventions: Drug: BI 3032950
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 3032950 — BI 3032950
  Arms: BI 3032950 treatment group - part A; BI 3032950 treatment group - part B
Drug: Placebo — Placebo
  Arms: Placebo group

SUMMARY:
The main objectives of this trial are to investigate safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of BI 3032950 in healthy male subjects following intravenous (Part A) or subcutaneous (Part B) administration of single rising doses.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 65 years (inclusive)
* BMI of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial
* Male subject (including male subjects with pregnant partners), who meets any of the following criteria for a highly effective contraception from at least timepoint of administration of trial medication until completion of end of trial (EoTrial) visit:

  * Use of combined (estrogen and progestogen containing) hormonal contraception that prevents ovulation (oral, intravaginal or transdermal) by female women of childbearing potential (WOCBP) partner, plus condom in male subject
  * Use of progestogen-only hormonal contraception that inhibits ovulation (only injectables or implants) by female WOCBP partner, plus condom in male subject
  * Use of intrauterine device (IUD) or intrauterine hormone-releasing system (IUS) by female WOCBP partner, plus condom in male subject
  * Male subject is sexually abstinent
  * Male subject is vasectomised (vasectomy at least 1 year prior to enrolment) and received medical assessment of the surgical success (documented absence of sperm)
  * Female partner is surgically sterilised (including hysterectomy, bilateral salpingectomy and bilateral oophorectomy)
  * Female partner is postmenopausal, defined as no menses for at least 1 year without an alternative medical cause (in questionable cases a blood sample with follicle stimulating hormone (FSH) above 40 U/L and estradiol below 30 ng/L is confirmatory, if available) Subjects are required to use condoms to prevent unintended exposure of their partner (both, male and female) to the trial drug via seminal fluid and should therefore use a condom at least from time point of administration of trial medication until completion of EoTrial visit. Alternatively, true abstinence is acceptable, if it is in line with the subject's preferred and usual lifestyle. If a subject is usually not sexually active, but becomes active with their partner, they must comply with the contraceptive requirements detailed above. Subjects should not donate sperm for the duration of the trial until completion of EoTrial visit.

Exclusion Criteria:

* Any finding in the medical examination (including blood pressure (BP), pulse rate (PR) or electrocardiogram (ECG)) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 100 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Relevant chronic or acute infections (including COVID-19 and active or latent tuberculosis)
* Further exclusion criteria apply

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2023-09-21 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with treatment-emergent adverse event | Up to 116 days

SECONDARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | Up to 113 days
Maximum measured concentration of the analyte in plasma (Cmax) | Up to 113 days
Percentage of subjects treated with investigational drug who experience a treatment emergent adverse event assessed as drug-related by the investigator | Up to 116 days

CONTACTS AND LOCATIONS:
Locations (1):
- SGS Life Science Services - Clinical Research, Edegem, Belgium

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com